CLINICAL TRIAL: NCT04356443
Title: Non-Invasive Monitoring of Respiratory Function in Spontaneously Breathing Patients With COVID-19 Infection
Status: Terminated | Type: Observational
Why Stopped: Technical challenges
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Omar Hyder, Anesthesia & Critical Care Attending Physician, Massachusetts General Hospital
Other Study IDs: 2020P000881
Record Dates: First submitted 2020-04-16; First posted 2020-04-22 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Respiratory Failure; Ventilatory Failure; COVID-19; Pneumonia; ARDS, Human
MeSH Terms: conditions — Respiratory Insufficiency; Hypoventilation; COVID-19; Pneumonia; Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

INTERVENTIONS:
Device: AirGo Respiratory Monitor — AirGo™ is composed of a wearable, miniaturized recorder unit and a medical grade Holter worn over the floating ribs of patients both at rest and during normal activity. The recorder measures live circumference changes.

SUMMARY:
This study uses the AirGo band to monitor changes in tidal ventilation in spontaneously breathing patients with COVID-19 associated respiratory failure. It aims to recognize patterns of ventilation associated with worsening respiratory failure in this patient population. If successful, this study will lead to the development of new robust methods for real-time, continuous monitoring of respiratory function in patients with respiratory failure. In turn, such monitoring methods may enable improvements in the medical management of respiratory failure and timing of interventions.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to the hospital
* ≥ 18 years of age
* Clinically suspected or confirmed COVID-19 infection
* Spontaneously breathing
* For patients not on supplemental oxygen at their location of residence prior to hospital admission, need for supplemental O2 to maintain SpO2 >=92%
* For patients on supplemental O2 at their location of residence prior to hospital admission, an increase in requirement of supplemental oxygen from baseline

Exclusion Criteria:

* Intubated patients
* Pregnant women
* Moribund patients
* Patients who are on comfort measures (CMO)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a pilot study that aims to recruit 500 patients with respiratory failure due to COVID-19 infection at Massachusetts General Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2020-04-15 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Endotracheal intubation during present hospitalization, recorded through chart review | Up to three weeks
  Progression of respiratory failure to require endotracheal intubation (and mechanical ventilation)

SECONDARY OUTCOMES:
Improvement in hypoxemia as indicated by oxygen saturation and requirement for supplemental oxygen, recorded through chart review | Up to three weeks
  Maintenance of SpO2 >=90% on no or low flow supplemental oxygen (=< 1 liter by nasal cannula or CPAP, or return of supplemental oxygen to baseline if required supplemental O2 for another indication, prior to onset of COVID-19 infection)
Premature need for removal of the band, recorded through investigator report | Up to three weeks
  Patient or care provider may request removal of the band for any reason prior to the patient reaching the outcome
In-hospital mortality, recorded through chart review | Up to 24 weeks
  Death from any cause while in the hospital

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No